CLINICAL TRIAL: NCT00149773
Title: Cognitive Therapy for Suicidal Older Men in Primary Care Settings
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P20MH071905-01 (NIH); P20MH071905-01 (NIH); 802223; DSIR 83-ATP
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2006-06

CONDITIONS: Suicide, Attempted
Keywords: Cognitive therapy; Suicide; Older men; Death ideation; Primary care
MeSH Terms: conditions — Suicide, Attempted; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Cognitive Therapy + Enriched Usual Care (Experimental): The cognitive therapy intervention consists of approximately 12 (1-hour) sessions over the course of a 4-month period. The main therapy components include:
  1. Using problem-solving and cognitive restructuring techniques to target hopelessness, reasons for living and dying, coping with loss, and perceived medical comorbidity that lead to suicidal ideation.
  2. Improving social resources.
  3. Improving adherence to medical regimen.
  4. Targeting Suicidal Cognitions.
  Interventions: Behavioral: Cognitive Therapy
- EnrichedUsual Care Condition (No Intervention): The Enriched Care (EC) condition will be used as the treatment comparison for this study. EC consists of usual care patients may obtain in the community as well as the assessment and referral services provided by the study case managers. Participation in the study does not restrict patients in any way in their access to other health care, and all patients in both conditions will be allowed to receive any additional mental health treatment in the community.
  The primary role of the study case manager is to establish a strong relationship with patients in order to retain the patients in the study for the duration of the study period.

INTERVENTIONS:
Behavioral: Cognitive Therapy
  Arms: Cognitive Therapy + Enriched Usual Care

SUMMARY:
This study will assess the effectiveness of cognitive therapy in reducing the incidence of suicide ideation and behavior in older men in a primary care setting.

DETAILED DESCRIPTION:
Older adult males have the highest suicide rate of any age group in the U.S. Over 70 percent of older suicide victims have been to their primary care physician within a month of their death, many with a depressive illness that was not detected. However, most research concerning treatments for suicide ideation and behavior has focused on adolescents and young adults. Very few treatments have been developed to reduce suicide ideation and behavior in men aged 60 and above. This study will assess the effectiveness of specialized cognitive therapy versus typical treatment in treating older men with suicide ideation.

Participants in this two-year, single-blind study will be randomly assigned to receive either cognitive therapy combined with enriched care or enriched care alone. Participants will be identified in primary care settings as having experienced suicide ideation in the past month. Cognitive therapy will be provided by Ph.D.-level therapists and will be geared specifically toward older men with suicidal tendencies. The enriched care condition will consist of the usual care that individuals receive for suicide prevention, plus assessment and referral services provided by independent evaluators and study case managers. All participants will be assessed pre-treatment to attain baseline measures of suicide ideation, hopelessness, and depression. Study visits will occur at baseline and Months 1, 3, 6, 12, 18, and 24 to assess suicide ideation. Self-report and clinician-administered measures will be used to assess participants' progress.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00218725

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing death ideation or suicidal ideation (total score greater than 0 on the Scale for Suicide Ideation)
* English-speaking
* Lives within the area served by the research unit
* Able to provide at least 2 verifiable contacts (typically family members)

Exclusion Criteria:

* Requires priority treatment for an acute, unstable, or severe Axis III disorder (e.g., dementia)
* Requires priority treatment for another debilitating problem (e.g., severe alcohol or drug dependence, mania, severe anorexia)
* Suffers from a psychotic disorder or psychotic thought processes
* Exhibits self-mutilating behavior without any intent to commit suicide (e.g., burning oneself with a cigarette)

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation; measured at Months 1, 3, 6, 12, 18, and 24 | 1, 3, 6, 12, 18, and 24 months

SECONDARY OUTCOMES:
Depression; measured at Months 1, 3, 6, 12, 18, and 24 | 1, 3, 6, 12, 18, and 24 months
Hopelessness; measured at Months 1, 3, 6, 12, 18, and 24 | 1, 3, 6, 12, 18, and 24 months
Perceived Social Support; measured at Months 1, 3, 6, 12, 18, and 24 | 1, 3, 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Aaron T. Beck, MD, Principal Investigator — University of Pennsylvania; Gregory K. Brown, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Psychopathology Research Unit - University of Pennsylvania, Philadelphia, Pennsylvania, United States